CLINICAL TRIAL: NCT03056313
Title: The Proactive Support of Labor Study
Acronym: PAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014/1788
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Obstetric Labor Complications
Keywords: Delivery, Obstetric; Uterine Contraction; Cervix Uteri
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proactive support of labor (Experimental): delayed labor; 1 cm opening and painful contractions
  Interventions: Behavioral: Proactive support of labor
- support of labor as usual (Active Comparator): delayed labor; 3-4 cm opening of the cervix and regular contractions
  Interventions: Behavioral: support of labor as usual

INTERVENTIONS:
Behavioral: Proactive support of labor — In case of delayed labor, active labor is defined at an earlier stage; labor support is given with 1 cm opening of the cervix and painful contractions. Labor support interventions are started then.
  Arms: proactive support of labor
Behavioral: support of labor as usual — In case of delayed labor, active labor start is defined as usual at 3-4 cm opening of the cervix and regular contractions. Labor support interventions are started then.
  Arms: support of labor as usual

SUMMARY:
The duration of labor is decisive for maternal and fetal health. Poor progression often results in tired mothers, bad experience, delivery complications and a demand for cesarean section in next pregnancy. Proactive support of labor is a method originally from the Netherlands.

The main idea is to define start of active labor earlier than the traditional "3-4 cm opening of the cervix and regular contractions" to be cervix < 0.5 cm in length, and 1 cm opening and painful contractions. From this point, it is expected to be a progress of 1cm/hour opening of cervix. If not, progress is supported by amniotomy or stimulation of contractions.

This method is embraced by several clinics with great enthusiasm. However, there are no randomized controlled trials to prove that this method is better than others.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous start of labor
* nulliparous
* term pregnancy
* cephalic presentation

Exclusion Criteria:

* twins
* breech presentation
* given birth earlier
* known uterine anomaly
* insulin treated diabetes
* preeclampsia
* other serious medical conditions in mother or fetus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 347 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
number of pathological deliveries | 2 days
  number non-normal deliveries
maternal satisfaction with deliver | 1 week
  validated Childbirth Experience Questionnaire (CEQ) (Anna Dencker 2010)

CONTACTS AND LOCATIONS:
Overall Officials: Eszter Vanky, md prof, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Background] Brenne Fehn M, Dahlo R, Nielsen R, Laache I, Vanky E. Proactive versus standard support of labour in nulliparous women; study protocol for a randomized, controlled trial. Trials. 2020 Apr 23;21(1):358. doi: 10.1186/s13063-020-4191-9. PMID 32326956